CLINICAL TRIAL: NCT02707276
Title: Low Field Magnetic Stimulation: Initial Trial in Geriatric Bipolar Depression
Brief Title: LFMS: Initial Trial in Geriatric Bipolar Depression
Acronym: LFMS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Limited resources and funding resulted in a decision to prematurely halt study and redirect remaining funds to partner study Low Field Magnetic Stimulation: Imaging Biomarkers in Geriatric Bipolar Depression (Protocol #2017P002783).
Sponsor: Mclean Hospital (Other)
Responsible Party: Principal Investigator, Brent Forester, Clinical Director, Mclean Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2015P001851
Record Dates: First submitted 2016-03-04; First posted 2016-03-14 (Estimated); Results first posted 2022-03-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-01

CONDITIONS: Bipolar Depression Depressed Phase
Keywords: Bipolar Depression; Geriatric; Low Field Magnetic Stimulation
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Intervention Model Description: There are two phases. The first, pilot phase was a randomized, double-blinded crossover design. Following review of data from a different Low Field Magnetic Stimulation study (2012P002380) that showed a large order effect from the crossover design, revision of study design was prompted. The study design for this second phase was a randomized, double-blinded sham-controlled parallel design.
Who Masked: Participant, Investigator
Masking Description: The system can operate in sham mode, with identical sounds to active mode. The system can be programmed to randomize subjects automatically without the knowledge of study staff.
Oversight: Data Monitoring Committee: No

ARMS (4):
- Phase 1: Cross-Over, Active LFMS first (Experimental): Phase 1 crossover: three 20 minute treatments of active low field magnetic stimulation, once per day for three consecutive days during week 1. Then repeat with three 20 minute treatments of sham LFMS, once per day for three consecutive days during week 3.
  Interventions: Device: Active Low Field Magnetic Stimulation
- Phase 1: Cross-Over, Sham LFMS first (Sham Comparator): Phase 1 crossover: three 20 minute treatments of sham low field magnetic stimulation, once per day for three consecutive days during week 1. Then repeat with three 20 minute treatments of active LFMS, once per day for three consecutive days during week 3.
  Interventions: Device: Sham Low Field Magnetic Stimulation
- Phase 2: Parallel, Active LFMS (Experimental): Phase 2 parallel: five 20-minute active low field magnetic stimulation treatments, once per day for five consecutive days during week 1.
  Interventions: Device: Active Low Field Magnetic Stimulation
- Phase 2: Parallel, Sham LFMS (Sham Comparator): Phase 2 parallel: five 20-minute sham low field magnetic stimulation treatments, once per day for five consecutive days during week 1.
  Interventions: Device: Sham Low Field Magnetic Stimulation

INTERVENTIONS:
Device: Active Low Field Magnetic Stimulation — Low Field Magnetic Stimulation is an electromagnetic treatment being investigated for its effects on mood. It uses magnetic fields that are a fraction of the strength but at a higher frequency than the electromagnetic fields used in transcranial magnetic stimulation (TMS) and electroconvulsive therapy (ECT)
  Other Names: Active LFMS
  Arms: Phase 1: Cross-Over, Active LFMS first; Phase 2: Parallel, Active LFMS
Device: Sham Low Field Magnetic Stimulation — The sham treatment does not provide any electromagnetic stimulation. However, it is designed so that it cannot be differentiated from the active treatment by producing mimicking sounds.
  Other Names: Sham LFMS
  Arms: Phase 1: Cross-Over, Sham LFMS first; Phase 2: Parallel, Sham LFMS

SUMMARY:
The primary aim of this study is to assess the efficacy of Low Field Magnetic Stimulation (LFMS) in treating symptoms of depression and anxiety in older adults suffering from bipolar depression. The investigators also aim to assess any cognitive benefits from regular LFMS treatments in older adults suffering from bipolar depression.

DETAILED DESCRIPTION:
The investigators have previously observed mood improvement in participants with bipolar depression in a population aged 21-60. Here the investigators hope to extend these results to a similar but new population, geriatric bipolar depression (GPD). In addition to the evaluation of the effect of multiple treatments, as well as observation of the duration of the effect after a delay of one week in this population, the investigators will assess whether this population presents any noticeable difference in tolerance or effect.

This study was completed in two phases; the design of the second phase was revised based on results from a related study (2012P002380). The first phase had a randomized, double-blind, sham-controlled crossover design. Subjects were distributed equally into two groups; one group received three active LFMS sessions during a first treatment week and three sham LFMS sessions during a second treatment week, while the second group received sham LFMS first and then active LFMS. Specifically, all subjects made a baseline visit during week 0 (visit 1, any day) where scales of depression (Montgomery-Asberg Rating Scale (MADRS)), anxiety (Hamilton Anxiety Rating Scale (HARS)), and positive affect (Positive and Negative Affect Schedule (PANAS)) were completed. Subjects returned during week 1 for three treatment visits (visits 2,3,4 any days) during which they received active or sham LFMS according to their order assignment. Subject returned for the same mood ratings during week 2 (visit 5, any day). Subjects returned during week 3 for three treatment visits and received the alternate treatment according to their order assignment (visits 6,7,8, any days). Finally, subjects returned week 4 for to receive the mood ratings (visit 9, any day). The MADRS, HARS, and PANAS scales completed during weeks 0, 2, and 4 were the outcome measures. Treatment order assignments were randomized and balanced within blocks of 10 via a random number generator.

Following review of data from a different Low Field Magnetic Stimulation study (2012P002380), the study design was revised, and a second phase of this protocol resulted. This is a randomized, double-blind, sham-controlled study with a parallel design (subjects will either receive active treatment or sham treatment for all treatment sessions). Specifically, the MADRS, HARS, and PANAS were completed on baseline visit 1 (day 0, Friday); 5 treatment visits were made on days 3,4,5,6,7 (visits 2-6); a mood rating visit 7 was made on day 10. The MADRS, HARS, and PANAS scales completed during days 0 and 10 were the outcome measures. Treatment order assignments were randomized and balanced within blocks of 10 via a random number generator.

The mechanisms of depression in a geriatric population may differ from those in a younger population. Brain structures and connectivity have changed, and there is the increased risk of comorbid diagnoses such as dementia that might confound treatment and assessment. In this study the investigators hope to extend the findings of LFMS in the general population to directly address the treatment of bipolar depression in a geriatric population.

ELIGIBILITY:
Inclusion criteria:

1. Subjects will be men or women aged 55 years or older.
2. Subjects will have a diagnosis of Bipolar Disorder Type I or II, current episode depressed as measure by a MADRS ≥ 20.
3. Subjects must have failed at least one FDA approved treatment for bipolar depression before enrolling in this study. Failed treatment is defined as 8 weeks of treatment at standard dose (Selective Serotonin Reuptake Inhibitors (SSRI) , Selective Norepinephrine Reuptake Inhibitors (SNRI), mood stabilizer, or typical or atypical antipsychotic).
4. Subjects must be maintained on a stable dose of all psychotropic medications for a period of at least two weeks prior to screening.
5. Subjects must be capable of providing informed consent.

Exclusion criteria:

1. Subjects meeting Diagnostic Statistical Manual-IV-TR (DSM-IV-TR) criteria for any Axis I disorder other than Bipolar Disorder or an anxiety disorder (eg. Major Depressive Disorder, dementia).
2. Subject has an Mini Mental State Exam (MMSE) score ≤ 24.
3. Subject is pregnant or plans on becoming pregnant.
4. Subject has recent history (within 7 days of screening) of ECT or TMS treatment.
5. Subject has recent history of substance abuse (cannot meet DSM-IV-TR criteria for substance abuse, no significant drug abuse within last 3 months, no history of dependence in last year, no drug use within last month, other than marijuana use).
6. Subject has any contraindication for Magnetic Resonance Imaging (MRI) (i.e. Presence of a pacemaker, neurostimulator, or metal in head or neck).

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-09-07 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brent Forester, M.D. MSc., Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment spanned from 2017 to 2019. 30 subjects in total were screened, while 16 of those subjects enrolled in the study. All subjects were recruited through the Mass General Brigham Clinical Trials Portal or through referrals via our internal McLean "Successful Aging through Group Engagement" program.
Pre-assignment Details: Enrolled subjects underwent thorough screening procedures to determine diagnostic status. Two subjects did not meet diagnostic criteria and thus were not assigned to a group. One subject withdrew from the study due to personal reasons before being assigned to a group.
Groups:
- Cross-Over Phase; Active LFMS First: Active Low Field Magnetic Stimulation before Sham Low Field Magnetic Stimulation
  Phase 1 crossover: three 20 minute treatments of active LFMS, once per day for three consecutive days. Then repeat with three 20 minute treatments of sham LFMS, once per day for three consecutive days
  Active Low Field Magnetic Stimulation: Low Field Magnetic Stimulation is an electromagnetic treatment being investigated for its effects on mood. It uses magnetic fields that are a fraction of the strength but at a higher frequency than the electromagnetic fields used in transcranial magnetic stimulation (TMS) and electroconvulsive therapy (ECT)
  Sham Low Field Magnetic Stimulation: The sham treatment does not provide any electromagnetic stimulation. However, it is designed so that it cannot be differentiated from the active treatment.
- Cross-Over Phase; Sham LFMS First: Sham Low Field Magnetic Stimulation before Active Low Field Magnetic Stimulation
  Phase 1 crossover: three 20 minute treatments of active LFMS, once per day for three consecutive days. Then repeat with three 20 minute treatments of sham LFMS, once per day for three consecutive days
  Active Low Field Magnetic Stimulation: Low Field Magnetic Stimulation is an electromagnetic treatment being investigated for its effects on mood. It uses magnetic fields that are a fraction of the strength but at a higher frequency than the electromagnetic fields used in transcranial magnetic stimulation (TMS) and electroconvulsive therapy (ECT)
  Sham Low Field Magnetic Stimulation: The sham treatment does not provide any electromagnetic stimulation. However, it is designed so that it cannot be differentiated from the active treatment.
- Parallel Phase; Active LFMS: Phase 2 parallel: five 20 minute treatments, once per day for five consecutive days
  Active Low Field Magnetic Stimulation: Low Field Magnetic Stimulation is an electromagnetic treatment being investigated for its effects on mood. It uses magnetic fields that are a fraction of the strength but at a higher frequency than the electromagnetic fields used in transcranial magnetic stimulation (TMS) and electroconvulsive therapy (ECT)
- Parallel Phase; Sham LFMS: Phase 2 parallel: five 20 minute treatments, once per day for five consecutive days
  Sham Low Field Magnetic Stimulation: The sham treatment does not provide any electromagnetic stimulation. However, it is designed so that it cannot be differentiated from the active treatment.
Period: Overall Study
Arm/Group | Cross-Over Phase; Active LFMS First | Cross-Over Phase; Sham LFMS First | Parallel Phase; Active LFMS | Parallel Phase; Sham LFMS
Started | 3 | 5 | 3 | 2
Completed | 3 | 5 | 3 | 2
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis population is the same as the assignment in the Participant Flow.
Groups:
- Phase 1: Cross-Over, Active LFMS First: Active Low Field Magnetic Stimulation before Sham Low Field Magnetic Stimulation
  Phase 1 crossover: three 20 minute treatments of active LFMS, once per day for three consecutive days. Then repeat with three 20 minute treatments of sham LFMS, once per day for three consecutive days
  Active Low Field Magnetic Stimulation: Low Field Magnetic Stimulation is an electromagnetic treatment being investigated for its effects on mood. It uses magnetic fields that are a fraction of the strength but at a higher frequency than the electromagnetic fields used in transcranial magnetic stimulation (TMS) and electroconvulsive therapy (ECT)
  Sham Low Field Magnetic Stimulation: The sham treatment does not provide any electromagnetic stimulation. However, it is designed so that it cannot be differentiated from the active treatment.
- Phase 1: Cross-Over, Sham LFMS First: Sham Low Field Magnetic Stimulation before Active Low Field Magnetic Stimulation
  Phase 1 crossover: three 20 minute treatments of active LFMS, once per day for three consecutive days. Then repeat with three 20 minute treatments of sham LFMS, once per day for three consecutive days
  Active Low Field Magnetic Stimulation: Low Field Magnetic Stimulation is an electromagnetic treatment being investigated for its effects on mood. It uses magnetic fields that are a fraction of the strength but at a higher frequency than the electromagnetic fields used in transcranial magnetic stimulation (TMS) and electroconvulsive therapy (ECT)
  Sham Low Field Magnetic Stimulation: The sham treatment does not provide any electromagnetic stimulation. However, it is designed so that it cannot be differentiated from the active treatment.
- Phase 2: Parallel, Active LFMS: Phase 2 parallel: five 20 minute treatments, once per day for five consecutive days
  Active Low Field Magnetic Stimulation: Low Field Magnetic Stimulation is an electromagnetic treatment being investigated for its effects on mood. It uses magnetic fields that are a fraction of the strength but at a higher frequency than the electromagnetic fields used in transcranial magnetic stimulation (TMS) and electroconvulsive therapy (ECT)
- Phase 2: Parallel, Sham LFMS: Phase 2 parallel: five 20 minute treatments, once per day for five consecutive days
  Sham Low Field Magnetic Stimulation: The sham treatment does not provide any electromagnetic stimulation. However, it is designed so that it cannot be differentiated from the active treatment.
- Total: Total of all reporting groups
Arm/Group | Phase 1: Cross-Over, Active LFMS First | Phase 1: Cross-Over, Sham LFMS First | Phase 2: Parallel, Active LFMS | Phase 2: Parallel, Sham LFMS | Total
Number analyzed (Participants) | 3 | 5 | 3 | 2 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.0 (5.2) | 66.4 (3.8) | 62.3 (11.0) | 71.5 (2.1) | 64.8 (6.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 2 | 1 | 7
  Male | 1 | 3 | 1 | 1 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 5 | 3 | 2 | 13
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 3 | 5 | 3 | 2 | 13
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
MADRS Baseline [Mean (Standard Deviation); unit: scores on a scale] — The Montgomery-Asberg Depression Rating Scale (MADRS) is a diagnostic assessment measuring the severity of depressive symptoms. It is a 10-item scale assessing all core symptoms of repression. Each item is scored on a 7-point scale, ranging from 0 (symptom not present) to 6 (symptom severely present). Thus, the total score range is 0-60, with higher scores indicating more depressive symptom endorsement.
  scores on a scale | 30.3 (7.02) | 25.4 (4.10) | 27.33 (11.93) | 22.5 (3.54) | 26.53 (6.75)
HARS Hamilton Anxiety Rating Scale [Mean (Standard Deviation); unit: scores on a scale] — The Hamilton Anxiety Rating Scale (HARS) assesses the severity of anxiety symptoms. It is a 14-item scale covering psychic and somatic anxiety. Each item is scored on a 5-point scale, ranging from 0 (not present) to 4 (severe). Thus, the total score range is 0-56, wither higher scores indicating higher anxiety severity.
  scores on a scale | 17.67 (7.77) | 12.4 (5.77) | 15.67 (4.93) | 13 (4.24) | 14.46 (5.64)
PANAS: Positive and Negative Affect Scale, Positive Subscale [Mean (Standard Deviation); unit: score on a scale] — The Positive and Negative Affect Schedule (PANAS) assesses the presence and severity of two factors: positive affect (PA) and negative affect (NA). The PANAS is a 20-item scale, with 10 items measured PA and 10 items measuring NA. Each item is scored on a 5-point scale ranging from 1 (very slightly/not at all) to 5 (extremely). The score range for PA is 10-50, and the score range for NA is 10-50, with higher scores indicated more endorsement of PA (more energy, concentration, and pleasure) or NA (more anger, disgust, contempt). This study reports data on the score ranges for the PA sub-scale.
  score on a scale | 20.33 (3.79) | 22.4 (11.28) | 25 (8.89) | 23.5 (9.19) | 22.69 (8.24)

OUTCOME MEASURES:

1. Primary Outcome: Change in Montgomery Asberg Depression Rating Scale (MADRS)
Description: The Montgomery-Asberg Depression Rating Scale (MADRS) is a diagnostic assessment measuring the severity of depressive symptoms. It is a 10-item scale assessing all core symptoms of repression. Each item is scored on a 7-point scale, ranging from 0 (symptom not present) to 6 (symptom severely present). Thus, the total score range is 0-60, with higher scores indicating more depressive symptom endorsement.
Time Frame: Phase 1 cross-over: scores at base visit 1 (week 0), visit 5 (week 2), and visit 9 (week 4). Differences are between visits 5-1 and 9-5. Phase 2 parallel: scores at base visit 1 (day 0) and visit 7 (day 10). Differences are between visits 7-1.
Measure: Mean (Standard Deviation); unit: score on scale
Groups:
- Phase 1: Cross-Over, Active LFMS First: Active Low Field Magnetic Stimulation
  Phase 1 crossover: three 20 minute treatments of active LFMS, once per day for three consecutive days. Then repeat with three 20 minute treatments of sham LFMS, once per day for three consecutive days
  Active Low Field Magnetic Stimulation: Low Field Magnetic Stimulation is an electromagnetic treatment being investigated for its effects on mood. It uses magnetic fields that are a fraction of the strength but at a higher frequency than the electromagnetic fields used in transcranial magnetic stimulation (TMS) and electroconvulsive therapy (ECT)
  Sham Low Field Magnetic Stimulation: The sham treatment does not provide any electromagnetic stimulation. However, it is designed so that it cannot be differentiated from the active treatment.
- Phase 1: Cross-Over, Sham LFMS First: Sham Low Field Magnetic Stimulation
  Phase 1 crossover: three 20 minute treatments of active LFMS, once per day for three consecutive days. Then repeat with three 20 minute treatments of sham LFMS, once per day for three consecutive days
  Active Low Field Magnetic Stimulation: Low Field Magnetic Stimulation is an electromagnetic treatment being investigated for its effects on mood. It uses magnetic fields that are a fraction of the strength but at a higher frequency than the electromagnetic fields used in transcranial magnetic stimulation (TMS) and electroconvulsive therapy (ECT)
  Sham Low Field Magnetic Stimulation: The sham treatment does not provide any electromagnetic stimulation. However, it is designed so that it cannot be differentiated from the active treatment.
Arm/Group | Phase 1: Cross-Over, Active LFMS First | Phase 1: Cross-Over, Sham LFMS First | Phase 2: Parallel, Active LFMS | Phase 2: Parallel, Sham LFMS
Number analyzed (Participants) | 3 | 5 | 3 | 2
score on scale
  Active LFMS | -13 (10.44) | 2.4 (14.15) | -7.67 (4.51) | NA (NA) — The Parallel Phase subjects were assigned to either active or sham LFMS groups, so they have no data to report in the rows which they did not participate in.
  Sham LFMS | 4.67 (5.86) | -7.2 (8.02) | NA (NA) — The Parallel Phase subjects were assigned to either active or sham LFMS groups, so they have no data to report in the rows which they did not participate in. | -2.50 (2.12)
Statistical Analysis 1: Comparison: Phase 1: Cross-Over, Active LFMS First vs Phase 1: Cross-Over, Sham LFMS First; Repeated measures ANCOVA with baseline MADRS scores as covariate for treatment and order effects of difference in MADRS scores; Test type: Superiority; p < 0.76, ANCOVA; repeated measures ANCOVA; Mean Difference (Final Values) = -0.625, Standard Deviation 12.0 — mean raw change active-sham; pooled standard deviation
Statistical Analysis 2: Comparison: Phase 2: Parallel, Active LFMS vs Phase 2: Parallel, Sham LFMS; ANCOVA: Analysis of group differences in change scores with baseline as a covariate; Test type: Superiority; p < 0.33, ANCOVA; Baseline covariate; Mean Difference (Final Values) = -5.17, Standard Deviation 4.96 — Pooled deviation

2. Primary Outcome: Change in Hamilton Anxiety Rating Scale (HARS)
Description: The Hamilton Anxiety Rating Scale (HARS) assesses the severity of anxiety symptoms. It is a 14-item scale covering psychic and somatic anxiety. Each item is scored on a 5-point scale, ranging from 0 (not present) to 4 (severe). Thus, the total score range is 0-56, wither higher scores indicating higher anxiety severity.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Phase 1: Cross-Over, Active LFMS First | Phase 1: Cross-Over, Sham LFMS First | Phase 2: Parallel, Active LFMS | Phase 2: Parallel, Sham LFMS
Number analyzed (Participants) | 3 | 5 | 3 | 2
score on a scale
  Active | -7.67 (10.69) | 4.2 (9.58) | 15.67 (4.93) | NA (NA) — The Parallel Phase subjects were assigned to either active or sham LFMS groups, so they have no data to report in the rows which they did not participate in.
  Sham | 3 (5.20) | -5.4 (5.32) | NA (NA) — The Parallel Phase subjects were assigned to either active or sham LFMS groups, so they have no data to report in the rows which they did not participate in. | -7.33 (3.214)
Statistical Analysis 1: Comparison: Phase 1: Cross-Over, Active LFMS First vs Phase 1: Cross-Over, Sham LFMS First; Repeated measures ANCOVA with baseline HARS scores as covariate for treatment and order effects of difference in HARS scores; Test type: Superiority; p < 0.61, ANCOVA; repeated measures ANCOVA; Mean Difference (Net) = 2.0, Standard Deviation 9.1 — raw change active-sham mean; pooled standard deviation
Statistical Analysis 2: Comparison: Phase 2: Parallel, Active LFMS vs Phase 2: Parallel, Sham LFMS; ANCOVA: Analysis of group differences in change scores with baseline as a covariate; Test type: Superiority; p < 0.32, ANCOVA; baseline as covariate; Mean Difference (Final Values) = -4.33, Standard Deviation 4.00 — pooled deviation

3. Primary Outcome: Change in Positive and Negative Affect Schedule (PANAS), Positive Sub Scale
Description: The Positive and Negative Affect Schedule (PANAS) assesses the presence and severity of two factors: positive affect (PA), which indicates the extent that a person is experiencing high energy, enthusiastic, mood state, and negative affect (NA), which indicates the extent a person is experiencing an aversive mood state. The PANAS is a 20-item scale, with 10 items measured PA and 10 items measuring NA. Each item is scored on a 5-point scale ranging from 1 (very slightly or not at all) to 5 (extremely). Thus, the score range for PA is 10-50, and the score range for NA is 10-50, with higher scores indicated more endorsement of PA (more energy, concentration, and pleasure) or NA (more anger, disgust, contempt). This study reports data on the score ranges for the PA sub-scale.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Phase 1: Cross-Over, Active LFMS First | Phase 1: Cross-Over, Sham LFMS First | Phase 2: Parallel, Active LFMS | Phase 2: Parallel, Sham LFMS
Number analyzed (Participants) | 3 | 5 | 3 | 2
score on a scale
  Active LFMS | -3 (7.2) | 1.2 (15.5) | -4.33 (4.16) | NA (NA) — The Parallel Phase subjects were assigned to either active or sham LFMS groups, so they have no data to report in the rows which they did not participate in.
  Sham LFMS | 4 (12.17) | -0.4 (2.45) | NA (NA) — The Parallel Phase subjects were assigned to either active or sham LFMS groups, so they have no data to report in the rows which they did not participate in. | -4 (2.83)
Statistical Analysis 1: Comparison: Phase 1: Cross-Over, Active LFMS First vs Phase 1: Cross-Over, Sham LFMS First; Repeated measures ANCOVA with baseline PANAS (Positive sub scale) scores as covariate for treatment and order effects of difference in PANAS (Positive sub scale) scores; Test type: Superiority; p < 0.78, ANCOVA; repeated measures ANCOVA; Mean Difference (Final Values) = -1.625, Standard Deviation 10.2 — raw active-sham mean; pooled standard deviation
Statistical Analysis 2: Comparison: Phase 2: Parallel, Active LFMS vs Phase 2: Parallel, Sham LFMS; ANCOVA: Analysis of group differences in change scores with baseline as a covariate; Test type: Superiority; p < 0.99, ANCOVA; baseline as covariate; Mean Difference (Final Values) = -0.33, Standard Deviation 2.42 — pooled deviation

ADVERSE EVENTS:
Time Frame: Participants in the cross-over phase were assessed over the course of 5 weeks, with the screen procedures occurring in week 1, active/sham treatments occurring in week 2, a follow-up in week 3, active/sham treatments occurring in week 4, and a follow-up in week 5. Participants in the parallel phase were assessed over the course of 4 weeks, with screening/baseline in week 1, five consecutive treatments in week 2, and one follow-up call per week for weeks 3 and 4.
Description: Definition of adverse event and/or serious adverse event was the same as the definition used by this website. Adverse events were queried for during every research visit.
Groups:
- Active LFMS: Includes subjects in phase 1 crossover: three 20 minute treatments of active LFMS, once per day for three consecutive days. Also includes subjects in parallel phase: five 20 minute treatments, once per day for five consecutive days.
  Active Low Field Magnetic Stimulation: Low Field Magnetic Stimulation is an electromagnetic treatment being investigated for its effects on mood. It uses magnetic fields that are a fraction of the strength but at a higher frequency than the electromagnetic fields used in transcranial magnetic stimulation (TMS) and electroconvulsive therapy (ECT)
- Sham LFMS: Includes subjects in phase 1 crossover: three 20 minute treatments of sham LFMS, once per day for three consecutive days. Also includes subjects in parallel phase: five 20 minute treatments, once per day for five consecutive days
  Sham Low Field Magnetic Stimulation: The sham treatment does not provide any electromagnetic stimulation. However, it is designed so that it cannot be differentiated from the active treatment.
Arm/Group | Active LFMS | Sham LFMS
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/7
Other Adverse Events (participants affected / at risk) | 2/6 | 2/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active LFMS (N=6) | Sham LFMS (N=7)
headache (Nervous system disorders) | 2 (2) | 1 (1) — headache that resolved spontaneously with cessation of treatment
Dizziness (Ear and labyrinth disorders) | 0 (0) | 1 (1) — Event resolved spontaneously with cessation of treatment
Pressure in Head (Nervous system disorders) | 0 (0) | 1 (1) — events resolve spontaneously with cessation of treatment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-17): https://cdn.clinicaltrials.gov/large-docs/76/NCT02707276/Prot_SAP_000.pdf